CLINICAL TRIAL: NCT05734391
Title: Surveillance of Healthcare-associated Infections & Antimicrobial Resistance
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Ebbing Lautenbach, Corrado Cancedda, University of Pennsylvania
Other Study IDs: 851492
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Antimicrobial Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal and rectal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- inpatients: Individuals in inpatient wards
  Interventions: Diagnostic Test: Routine Infection control

INTERVENTIONS:
Diagnostic Test: Routine Infection control — routine part of hospital IPC activities
  Other Names: Surveillance activity

SUMMARY:
The aims of this project, called "Surveillance of Healthcare-associated infections & Antimicrobial Resistance", or "SHARE", are to 1) enhance laboratory capacity to detect emerging AMR patterns; 2) strengthen hospital epidemiology programs to use data to prevent, detect, and contain emerging AMR threats; 3) deploy study teams to answer critical public health surveillance questions, and 4) to build a national network of infection prevention and control (IPC) resources to prevent, detect, and contain emerging infectious disease threats

DETAILED DESCRIPTION:
The World Health Organization (WHO) has declared antimicrobial resistance (AMR) one of the top 10 global public health threats facing humanity. AMR burden is higher in low-and-middle-income countries (LMICs) where, in recent decades, incidence and mortality from healthcare-associated infections (HAI) due to multidrug resistant organisms (MDRO) have dramatically increased. For example, neonatal sepsis is the third most common cause of neonatal deaths and multidrug-resistant Gram-negative bacteria are now the leading cause of sepsis among hospitalized neonates in south Asia and sub-Saharan Africa, including Botswana.1,2 One in three newborns with an MDRO bloodstream infection will die.3 In 2021, to respond to the global threat of AMR, U.S. Centers for Disease Control & Prevention (CDC) announced the launch of a global "network of networks" to tackle the problem of AMR and healthcare-associated infections (HAIs). The network, called "Global Antimicrobial Resistance Laboratory and Response Network", solicited funding applications; in December of 2021, Botswana was announced as recipient of a 5-year cooperative agreement following the successful application for funding for a comprehensive AMR surveillance project. The project was developed by investigators from Botswana-UPenn Partnership (BUP) in collaboration with Botswana's Ministry of Health & Wellness (MOHW) and the University of Botswana (UB).

ELIGIBILITY:
Inclusion Criteria:

* hospital inpatient admission to participating wards.

Exclusion Criteria:

* diagnosis of a bleeding disorder
* platelet counts of <50,000
* diagnosis of coagulopathy
* presence of active bleeding
* inability to have a nares swab collected due to some other condition where nasal swabbing would be contraindicated
* inability to have a rectal swab collected due to some other condition where rectal swabbing would be contraindicated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals being admitted to participating wards, of all clinical conditions, genders, and ages, meeting the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Expertise | 12 months
  Ultimately, the goal of the SHARE project is to assemble the expertise and infrastructure needed to build a resilient HAI/AMR surveillance system fully-incorporated into MOHW's surveillance activities. The project aims to build capacity, both material and knowledge, in existing laboratory and IPC teams to face the dynamic challenges posed by HAIs and AMR

SECONDARY OUTCOMES:
Feasibility and Surveillance | 12 months
  SHARE's "Colonization Feasibility Study", will seek to assess the feasibility and surveillance potential of routine MDRO screening in hospitals, determining whether MDRO colonization can provide an "early warning system" for emerging AMR threats

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD, MPH, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States
- Princess Marina Hospital, Gaborone, Botswana